CLINICAL TRIAL: NCT04413097
Title: Delayed Cord Clamping With Oxygen In Extremely Low Gestation Infants
Acronym: DOXIE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Sharp Mary Birch Hospital for Women & Newborns (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DOXIE; 5R03HD105224-02 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: IVH- Intraventricular Hemorrhage; Extreme Prematurity; Hypoxia Neonatal; Hyperoxia; Respiratory Insufficiency
Keywords: Delayed Cord Clamping; IVH- Intraventricular Hemorrhage; Hyperoxia in Neonates; Hypoxia Neonatal; Continuous Positive Airway Pressure (CPAP)
MeSH Terms: conditions — Asphyxia Neonatorum; Hyperoxia; Respiratory Insufficiency | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once consent is obtained and the research staff is notified of a subject's impending birth, our research team member will open a randomization card and set the oxygen blender on the special bed to either an FiO2 of .30 or 1.0 and cover the blender. The research team member will not be involved in the clinical care for the infant and will blind the clinical care team from the randomized assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCC and Low Oxygen Concentration (Active Comparator): During 90 seconds of delayed cord clamping, the infant will receive gentle stimulation and start CPAP by 30 seconds of life at an FiO2 .30, with CPAP of 5 cmH20. If the infant is apneic or there is no Pedicap color change the team will begin positive pressure ventilation (starting PIP of 20 cmH20) by 60 seconds of life. The infant will remain on this support up until the umbilical cord is clamped at 90 seconds or greater. Once the cord is clamped the infant resuscitation will continue according to unit protocol.
  Interventions: Procedure: Delayed Cord Clamping with Low Oxygen concentration
- DCC and High Oxygen Concentration (Experimental): During 90 seconds of delayed cord clamping, the infant will receive gentle stimulation and start CPAP by 30 seconds of life at an FiO2 1.0, with CPAP of 5 cmH20. If the infant is apneic or there is no Pedicap color change the team will begin positive pressure ventilation (starting PIP of 20 cmH20) by 60 seconds of life. The infant will remain on this support up until the umbilical cord is clamped at 90 seconds or greater. Once the cord is clamped the infant resuscitation will continue according to unit protocol.
  Interventions: Procedure: Delayed Cord Clamping with High Oxygen concentration

INTERVENTIONS:
Procedure: Delayed Cord Clamping with Low Oxygen concentration — During delayed umbilical cord clamping of 90 seconds, breathing assistance with CPAP/PPV and low oxygen concentration (FiO2 0.30) will be provided.
  Other Names: DCC with Low Oxygen concentration; DCC LO group
  Arms: DCC and Low Oxygen Concentration
Procedure: Delayed Cord Clamping with High Oxygen concentration — During delayed umbilical cord clamping of 90 seconds, breathing assistance with CPAP/PPV and high oxygen concentration (FiO2 1.0) will be provided.
  Other Names: DCC with High Oxygen concentration; DCC HI group
  Arms: DCC and High Oxygen Concentration

SUMMARY:
This study is being conducted to compare the incidence of preterm infants (up to 28+6 weeks GA) who achieve a peripheral oxygen saturation of 80 percent by 5 minutes of life (MOL) given mask CPAP/PPV with an FiO2 of 1.0 during DCC for 90 seconds (HI Group) to infants given mask CPAP/PPV with an FiO2 of .30 during DCC for 90 seconds (LO Group).

DETAILED DESCRIPTION:
Prenatal consent will be obtained on infant's with estimated gestational age up to 28+6 weeks. Shortly before delivery, infant's will be randomly assigned to receive either Low oxygen concentration (FiO2 .30) OR High oxygen concentration (FiO2 1.0) during 90 seconds of delayed cord clamping.

Randomization and intervention will remain blinded to the clinical care team during the entire study period. The research team member will open a randomization card when notified of a subject's impending birth, review the protocol with the obstetric provider performing the procedure, set-up the sterile stabilization bed, and note the time it takes from delivery until the clamping and cutting of the umbilical cord in both groups.

The research team member will set the oxygen blender as indicated by the randomization card and cover the blender to blind the FiO2 setting. The research team member will not be involved in the clinical care of the infant. The oxygen blender will be concealed from the clinical care team to ensure resuscitation maneuvers will not be biased.

Data will be submitted to the statistician, who will remain blinded to the intervention for the duration of the study.

At delivery, the infant will be placed on a platform that allows the infant to be close to the mother and the umbilical cord to remain intact for DCC. These beds are equipped with an oxygen blender, humidifier, t-piece resuscitator with mask, necessary to provide CPAP/PPV. At some centers the bed will be equipped with a radian warmer (Ceramotherm, Wyer GmbH, Germany) to maintain thermoregulation on the infant during delayed cord clamping.

If an infant is randomized to the DCC and Low Oxygen concentration (DCC LO group), the following procedure will ensue:

During delayed cord clamping, the infant will be gently stimulated by drying the infant with a sterile towel and provide CPAP by 30 seconds of life. During delayed cord clamping, breathing assistance with CPAP of 5 cm H20 and a FiO2 0.3 will be provided.

If an infant is randomized to the DCC and High Oxygen concentration (DCC HI group), the following procedure will ensue:

During delayed cord clamping, the infant will be gently stimulated by drying the infant with a sterile towel and provide CPAP by 30 seconds of life. During delayed cord clamping, breathing assistance with CPAP of 5 cm H20 and a FiO2 1.0 will be provided.

Patency of the airway in both groups will be assessed by a Colorimetric CO2 detector. Lack of color change will indicate that the airway is not patent (obstructed), the pressure is not sufficient to expand the lungs, there was excessive air leak, or there was no or inadequate pulmonary blood flow. If there is no color change, the neonatal provider will reposition and reattempt to open the airway, if no improvement they will initiate PPV (starting PIP of 20 cm H20) by 60 seconds of life. Cord clamping will occur at 90 seconds or greater and the infant will be transferred to a standard neonatal warmer and resuscitated per NRP guidelines.

Additionally, when available heart rate data will be collected using a non-invasive dry-electrode monitor, (NeoBeat, Laerdal Medical, Stavanger, Norway) and applied over the infant's chest or abdomen to provide continuous display of heart rate during 90 seconds of DCC.

Pulse oximetry, ECG sensors and Near-Infrared Spectroscopy (NIRS) sensors will be applied after cord clamping. The NIRS sensor will be placed on the infant's forehead. Cerebral StO2, SpO2, blood pressure (once in the NICU) and Heart rate will be recorded every two seconds and linked with other variables. These variables will continue to be recorded for the first 24 hours of life.

Blood sample will be collected at two different time points: Cord blood sample (T1: Cord blood collected after the cord is cut) and at 2 hours of life or NICU admission (T2). This is extra few drops of blood that is drawn from the baby for medical purposes (cord blood from cord gases and admission blood work up).

Samples will be tested for oxidized and reduced glutathione which are the most reliable and comprehensive biomarkers of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* up to 28+6 weeks Gestational age
* Single and Multiple pregnancy
* All modes of delivery (vaginally or caesarean section)

Exclusion Criteria:

* Parents decline consent
* Congenital anomalies of the newborn
* Bleeding Accreta
* Monochorionic multiples with evidence of TTTS
* Fetal or maternal risk (i.e. compromise)
* Preterm Premature Rupture of Membranes prior to 20 weeks gestation
* Parents request no resuscitation

Ages: 22 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of administration of oxygen during delayed cord clamping and it's impact on the incidence of preterm infants (up to 28 +6 weeks) who achieve a peripheral oxygen saturation of 80 percent by 5 minutes of life | by 5 minutes of life
  To assess the feasibility and compare the incidence of preterm infants (up to 28+6 weeks GA) who achieve a peripheral oxygen saturation of 80 percent by 5 MOL given mask CPAP/PPV with an FiO2 of 1.0 during DCC for 90 seconds (HI Group) to infants given mask CPAP/PPV with an FiO2 of .30 during DCC for 90 seconds (LO Group).

SECONDARY OUTCOMES:
All Grade IVH | Through study completion at hospital discharge, up to 6 months corrected gestational age (CGA)
  Any Intraventricular Hemorrhage (grades 1-4)
Frequency of Grade III and IV intraventricular hemorrhage | Through study completion at hospital discharge, up to 6 months corrected gestational age (CGA)
  Intraventricular hemorrhages (grades 3-4) (bleeding in the brain parenchyma and/or ventricular dilation
Resuscitation interventions | In the first 10 minutes of life
  Resuscitation interventions including intubation, chest compressions, medications
Changes in heart rate (BPM) in the first 10 minutes of life | In the first 10 minutes of life
  Changes in heart rate (BPM) in the first 10 minutes of life

OTHER OUTCOMES:
Changes in Inspired fractional oxygen (FiO2) | In the first 10 minutes of life
  Changes in Inspired fractional oxygen (FiO2)
Duration of Hypoxia | The first 10 minutes of life in the delivery room
  Duration of Hypoxia (defined as oxygen saturation<25th percentile of target ranges defined by Dawson et al.) in the first 10 minutes after birth
Duration of Hyperoxia | The first 10 minutes of life in the delivery room
  Duration of Hyperoxia (defined as oxygen saturation>95%) in the first 10 minutes after birth
Changes in Mean airway pressure, MAP (cm H20) | In the first 10 minutes of life
  Changes in Mean airway pressure, MAP (cm H20)
Duration of Positive Pressure Ventilation | The first 10 minutes of life in the delivery room
  Duration of positive pressure ventilation
Blood pressures in the first 24 hours of life | In the first 24 hours of life
  Blood pressures every hour in the first 24 hours of life
Cerebral tissue oxygenation in the first 24 hours of life | In the first 24 hours of life
  Cerebral tissue oxygenation in the first 24 hours of life
Average oxygen saturation in the first 5 minutes after birth | by 5 minutes of life
  Oxygen saturation in the first 5 minutes after birth
Average Heart rate in the first 5 minutes after birth | by 5 minutes of life
  Heart rate in the first 5 minutes after birth
Intubation in the Delivery room or Neonatal Intensive Care Unit (NICU) | Birth through study completion at discharge, up to 6 months of corrected gestational age
  Intubation in the Delivery room or Neonatal Intensive Care Unit (NICU)
Lowest and Highest Hemoglobin and/or Hematocrit | First 24 hours of life
  Hemoglobin and/or Hematocrit levels (before transfusion)
Mean arterial blood pressure | First 24 hours of life
  Mean arterial blood pressure (collected hourly)
Medication for Low Blood Pressure | First 24 hours of life
  Medication for Low Blood Pressure (e.g. hydrocortisone or pressors)
CRIB-II (Clinical Risk Index for Babies) | First 12 hours of life
  CRIB-II (Clinical Risk Index for Babies)
Duration of mechanical ventilation and/or CPAP | Birth through study completion at discharge, up to 6 months of corrected gestational age
  Number of days on mechanical ventilation and/or CPAP
Surfactant administration | Immediately after intervention through study completion at hospital discharge, up to 6 months of corrected gestational age
  Surfactant administration
Number of RBC Transfusions since birth | First 10 days after birth
  Number of RBC Transfusions since birth
Patent Ductus Arteriosus requiring pharmacological or surgical treatment | Through study completion at discharge, up to 6 months of corrected gestational age
  Patent Ductus Arteriosus requiring pharmacological or surgical treatment
Spontaneous Intestinal Perforation (SIP) requiring surgery or peritoneal drain | Through study completion at discharge, up to 6 months of corrected gestational age
  Spontaneous Intestinal Perforation (SIP) requiring surgery or peritoneal drain
Necrotizing Enterocolitis (Modified Bell's stage 2-3) | Through study completion at discharge, up to 6 months of corrected gestational age
  Necrotizing Enterocolitis (Modified Bell's stage 2-3)
Bronchopulmonary Dysplasia (mode of respiratory support administered at 36 weeks postmenstrual age; as defined and categorized in; Jensen, Dysart, Gantz, et al: Defining Bronchopulmonary Dysplasia) http://www.ncbi.nlm.nih.gov/pmc/articles/pmc6775872/ | Hospital course until 36 weeks PMA
  Bronchopulmonary Dysplasia (mode of respiratory support administered at 36 weeks postmenstrual age; as defined and categorized in; Jensen, Dysart, Gantz, et al: Defining Bronchopulmonary Dysplasia) http://www.ncbi.nlm.nih.gov/pmc/articles/pmc6775872/
Severe ROP (stage 3 or treated with laser or bevacizumab) | After the intervention through study completion at hospital discharge, up to 6 months of corrected gestational age
  Severe ROP (stage 3 or treated with laser or bevacizumab)
Combined outcome of severe IVH and/or death | Through study completion at death or discharge, up to 6 months of corrected gestational age
  Combined outcome of severe IVH and/or death
Death | Through study completion at death or discharge, up to 6 months of corrected gestational age
  Death
SVC Flow | 6 hours of life
  Superior Vena Cava flow by echocardiography
RVO | 6 hours of life
  Right Ventricular output by echocardiography
Left Ventricular Output | 6 hours of life
  Left Ventricular output by echocardiography
Cognitive Composite Score | 24 months corrected age
  Composite Score (cognitive 45-155; higher scores are better) as assessed by the Bayley Scales of Infant and Toddler Development Fourth Edition
Language Composite Score | 24 months corrected age
  Composite Score (language 45-155; higher scores are better) as assessed by the Bayley Scales of Infant and Toddler Development Fourth Edition
Motor Composite Score | 24 months corrected age
  Composite Score (motor 45-155; higher scores are better) as assessed by the Bayley Scales of Infant and Toddler Development Fourth Edition
Cerebral Palsy | 24 months corrected age
  As assessed by Gross Motor Function Classification System (GMFCS) Levels 1-5
Neurodevelopmental Outcome at 2 Years of Age | 22-26 months corrected age
  Overall and Domain Scores- Ages and Stages, 3rd ed. Questionnaire
Pulsatility Index | 6 hours of life
  Pulsatility index calculated from Doppler of the Middle Cerebral Artery
Resistive Index | 6 hours of life
  Resistive index calculated from Doppler of the Middle Cerebral Artery
Changes in cerebral oxygenation saturation, StO2 (%) | In the first 10 minutes of life
  Changes in cerebral oxygenation saturation, StO2 (%)
Changes in SpO2 (%) in the first 10 minutes of life | In the first 10 minutes of life
  Changes in SpO2 (%) in the first 10 minutes of life
Inhaled Nitric Oxide | Immediately after intervention through study completion at hospital discharge, up to 6 months of corrected gestational age
  Use of Inhaled Nitric Oxide for Respiratory failure or Pulmonary Hypertension
Glutathione (GSH/GSSG ratio) | from birth up to NICU admission or in the first 2 hours of life
  Assessment of oxidative biomarkers from birth up to 2 hours of life
Thermoregulation | from 5 minutes of life up to NICU admission in the first 2 hours of life
  Assessment of thermoregulation (axillary temperatures measured in degrees Celsius) during delayed cord clamping on extremely low gestational infants
Rate of Early Onset Sepsis | From birth up to 72 hours of life
  assessment of early onset sepsis with a positive blood or CSF culture at </= 72 HOL
Rate of Late Onset Sepsis | From > 72 hours of life through study completion at death or discharge, up to 6 months of corrected gestational age
  assessment of late onset sepsis with a positive blood or CSF culture at > 72 HOL

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - University of California Davis, Davis, California
  - University of California San Diego Jacobs Medical Center, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NICHD requirements (National Institute of Child Health and Human Development)
Supporting Information: SAP
Time Frame: 2 years after primary publication
Access Criteria: An archived dataset with documentation will be made available for additional users by outside investigators, in collaboration with the study investigators. We will work with NICHD program staff to develop a broad data sharing plan over time.

REFERENCES:
- [Background] Mercer JS, McGrath MM, Hensman A, Silver H, Oh W. Immediate and delayed cord clamping in infants born between 24 and 32 weeks: a pilot randomized controlled trial. J Perinatol. 2003 Sep;23(6):466-72. doi: 10.1038/sj.jp.7210970. PMID 13679933
- [Background] Rabe H, Jewison A, Fernandez Alvarez R, Crook D, Stilton D, Bradley R, Holden D; Brighton Perinatal Study Group. Milking compared with delayed cord clamping to increase placental transfusion in preterm neonates: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):205-211. doi: 10.1097/AOG.0b013e3181fe46ff. PMID 21252731
- [Background] Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. doi: 10.1542/peds.2005-1706. PMID 16585320
- [Background] Hofmeyr GJ, Bolton KD, Bowen DC, Govan JJ. Periventricular/intraventricular haemorrhage and umbilical cord clamping. Findings and hypothesis. S Afr Med J. 1988 Jan 23;73(2):104-6. PMID 3340910
- [Background] Hofmeyr GJ, Gobetz L, Bex PJ, Van der Griendt M, Nikodem C, Skapinker R, Delahunt T. Periventricular/intraventricular hemorrhage following early and delayed umbilical cord clamping. A randomized controlled trial. Online J Curr Clin Trials. 1993 Dec 29;Doc No 110:[2002 words; 26 paragraphs]. PMID 8305996
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. Early versus delayed umbilical cord clamping in preterm infants. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003248. doi: 10.1002/14651858.CD003248.pub2. PMID 15495045
- [Background] Fogarty M, Osborn DA, Askie L, Seidler AL, Hunter K, Lui K, Simes J, Tarnow-Mordi W. Delayed vs early umbilical cord clamping for preterm infants: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Jan;218(1):1-18. doi: 10.1016/j.ajog.2017.10.231. Epub 2017 Oct 30. PMID 29097178
- [Background] Wyllie J, Perlman JM, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e169-201. doi: 10.1016/j.resuscitation.2015.07.045. Epub 2015 Oct 15. No abstract available. PMID 26477424
- [Background] Polglase GR, Dawson JA, Kluckow M, Gill AW, Davis PG, Te Pas AB, Crossley KJ, McDougall A, Wallace EM, Hooper SB. Ventilation onset prior to umbilical cord clamping (physiological-based cord clamping) improves systemic and cerebral oxygenation in preterm lambs. PLoS One. 2015 Feb 17;10(2):e0117504. doi: 10.1371/journal.pone.0117504. eCollection 2015. PMID 25689406
- [Background] Hooper SB, Te Pas AB, Lang J, van Vonderen JJ, Roehr CC, Kluckow M, Gill AW, Wallace EM, Polglase GR. Cardiovascular transition at birth: a physiological sequence. Pediatr Res. 2015 May;77(5):608-14. doi: 10.1038/pr.2015.21. Epub 2015 Feb 4. PMID 25671807
- [Background] Bhatt S, Polglase GR, Wallace EM, Te Pas AB, Hooper SB. Ventilation before Umbilical Cord Clamping Improves the Physiological Transition at Birth. Front Pediatr. 2014 Oct 20;2:113. doi: 10.3389/fped.2014.00113. eCollection 2014. PMID 25368858
- [Background] Katheria A, Reister F, Essers J, Mendler M, Hummler H, Subramaniam A, Carlo W, Tita A, Truong G, Davis-Nelson S, Schmolzer G, Chari R, Kaempf J, Tomlinson M, Yanowitz T, Beck S, Simhan H, Dempsey E, O'Donoghue K, Bhat S, Hoffman M, Faksh A, Arnell K, Rich W, Finer N, Vaucher Y, Khanna P, Meyers M, Varner M, Allman P, Szychowski J, Cutter G. Association of Umbilical Cord Milking vs Delayed Umbilical Cord Clamping With Death or Severe Intraventricular Hemorrhage Among Preterm Infants. JAMA. 2019 Nov 19;322(19):1877-1886. doi: 10.1001/jama.2019.16004. PMID 31742630
- [Background] Katheria AC, Hassen K, Rich W, Poeltler D, Finer N. Resuscitation outcomes of infants that do not achieve a 5 min target SpO2 saturation. J Perinatol. 2019 Dec;39(12):1635-1639. doi: 10.1038/s41372-019-0491-x. Epub 2019 Sep 5. PMID 31488904
- [Background] Oei JL, Finer NN, Saugstad OD, Wright IM, Rabi Y, Tarnow-Mordi W, Rich W, Kapadia V, Rook D, Smyth JP, Lui K, Vento M. Outcomes of oxygen saturation targeting during delivery room stabilisation of preterm infants. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F446-F454. doi: 10.1136/archdischild-2016-312366. Epub 2017 Oct 7. PMID 28988158
- [Background] Katheria A, Poeltler D, Durham J, Steen J, Rich W, Arnell K, Maldonado M, Cousins L, Finer N. Neonatal Resuscitation with an Intact Cord: A Randomized Clinical Trial. J Pediatr. 2016 Nov;178:75-80.e3. doi: 10.1016/j.jpeds.2016.07.053. Epub 2016 Aug 26. PMID 27574999
- [Background] Duley L, Dorling J, Pushpa-Rajah A, Oddie SJ, Yoxall CW, Schoonakker B, Bradshaw L, Mitchell EJ, Fawke JA; Cord Pilot Trial Collaborative Group. Randomised trial of cord clamping and initial stabilisation at very preterm birth. Arch Dis Child Fetal Neonatal Ed. 2018 Jan;103(1):F6-F14. doi: 10.1136/archdischild-2016-312567. Epub 2017 Sep 18. PMID 28923985
- [Background] Dekker J, Martherus T, Lopriore E, Giera M, McGillick EV, Hutten J, van Leuteren RW, van Kaam AH, Hooper SB, Te Pas AB. The Effect of Initial High vs. Low FiO2 on Breathing Effort in Preterm Infants at Birth: A Randomized Controlled Trial. Front Pediatr. 2019 Dec 12;7:504. doi: 10.3389/fped.2019.00504. eCollection 2019. PMID 31921719
- [Background] Vaucher YE, Peralta-Carcelen M, Finer NN, Carlo WA, Gantz MG, Walsh MC, Laptook AR, Yoder BA, Faix RG, Das A, Schibler K, Rich W, Newman NS, Vohr BR, Yolton K, Heyne RJ, Wilson-Costello DE, Evans PW, Goldstein RF, Acarregui MJ, Adams-Chapman I, Pappas A, Hintz SR, Poindexter B, Dusick AM, McGowan EC, Ehrenkranz RA, Bodnar A, Bauer CR, Fuller J, O'Shea TM, Myers GJ, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network. Neurodevelopmental outcomes in the early CPAP and pulse oximetry trial. N Engl J Med. 2012 Dec 27;367(26):2495-504. doi: 10.1056/NEJMoa1208506. PMID 23268664
- [Background] Bhatt S, Alison BJ, Wallace EM, Crossley KJ, Gill AW, Kluckow M, te Pas AB, Morley CJ, Polglase GR, Hooper SB. Delaying cord clamping until ventilation onset improves cardiovascular function at birth in preterm lambs. J Physiol. 2013 Apr 15;591(8):2113-26. doi: 10.1113/jphysiol.2012.250084. Epub 2013 Feb 11. PMID 23401615
- [Background] Crawshaw JR, Kitchen MJ, Binder-Heschl C, Thio M, Wallace MJ, Kerr LT, Roehr CC, Lee KL, Buckley GA, Davis PG, Flemmer A, Te Pas AB, Hooper SB. Laryngeal closure impedes non-invasive ventilation at birth. Arch Dis Child Fetal Neonatal Ed. 2018 Mar;103(2):F112-F119. doi: 10.1136/archdischild-2017-312681. Epub 2017 Oct 20. PMID 29054974
- [Background] van Vonderen JJ, Hooper SB, Hummler HD, Lopriore E, te Pas AB. Effects of a sustained inflation in preterm infants at birth. J Pediatr. 2014 Nov;165(5):903-8.e1. doi: 10.1016/j.jpeds.2014.06.007. Epub 2014 Jul 16. PMID 25039041
- [Background] Davey MG, Moss TJ, McCrabb GJ, Harding R. Prematurity alters hypoxic and hypercapnic ventilatory responses in developing lambs. Respir Physiol. 1996 Aug;105(1-2):57-67. doi: 10.1016/0034-5687(96)00038-2. PMID 8897651
- [Background] Katheria AC, Brown MK, Faksh A, Hassen KO, Rich W, Lazarus D, Steen J, Daneshmand SS, Finer NN. Delayed Cord Clamping in Newborns Born at Term at Risk for Resuscitation: A Feasibility Randomized Clinical Trial. J Pediatr. 2017 Aug;187:313-317.e1. doi: 10.1016/j.jpeds.2017.04.033. Epub 2017 May 16. PMID 28526223
- [Background] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal Resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S204-41. doi: 10.1161/CIR.0000000000000276. No abstract available. PMID 26472855
- [Background] Vento M, Aguar M, Escobar J, Arduini A, Escrig R, Brugada M, Izquierdo I, Asensi MA, Sastre J, Saenz P, Gimeno A. Antenatal steroids and antioxidant enzyme activity in preterm infants: influence of gender and timing. Antioxid Redox Signal. 2009 Dec;11(12):2945-55. doi: 10.1089/ars.2009.2671. PMID 19645572
- [Background] Egan EA, Olver RE, Strang LB. Changes in non-electrolyte permeability of alveoli and the absorption of lung liquid at the start of breathing in the lamb. J Physiol. 1975 Jan;244(1):161-79. doi: 10.1113/jphysiol.1975.sp010789. PMID 1123740
- [Background] Walters DV, Olver RE. The role of catecholamines in lung liquid absorption at birth. Pediatr Res. 1978 Mar;12(3):239-42. doi: 10.1203/00006450-197803000-00017. PMID 205826
- [Background] Zhang Y, Chan GS, Tracy MB, Lee QY, Hinder M, Savkin AV, Lovell NH. Cerebral near-infrared spectroscopy analysis in preterm infants with intraventricular hemorrhage. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:1937-40. doi: 10.1109/IEMBS.2011.6090547. PMID 22254711
- [Background] Sorensen LC, Maroun LL, Borch K, Lou HC, Greisen G. Neonatal cerebral oxygenation is not linked to foetal vasculitis and predicts intraventricular haemorrhage in preterm infants. Acta Paediatr. 2008 Nov;97(11):1529-34. doi: 10.1111/j.1651-2227.2008.00970.x. Epub 2008 Jul 31. PMID 18673361
- [Background] Raju TN. Research in perinatal and neonatal medicine--a scientific vision for future decades. Indian J Pediatr. 2014 Jun;81(6):570-7. doi: 10.1007/s12098-014-1467-7. Epub 2014 May 14. PMID 24820234
- [Background] Fanaroff JM, Wilson-Costello DE, Newman NS, Montpetite MM, Fanaroff AA. Treated hypotension is associated with neonatal morbidity and hearing loss in extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1131-5. doi: 10.1542/peds.2005-1230. PMID 16585307
- [Background] Fanaroff AA, Fanaroff JM. Short- and long-term consequences of hypotension in ELBW infants. Semin Perinatol. 2006 Jun;30(3):151-5. doi: 10.1053/j.semperi.2006.04.006. PMID 16813974
- [Background] Laughon M, Bose C, Allred E, O'Shea TM, Van Marter LJ, Bednarek F, Leviton A; ELGAN Study Investigators. Factors associated with treatment for hypotension in extremely low gestational age newborns during the first postnatal week. Pediatrics. 2007 Feb;119(2):273-80. doi: 10.1542/peds.2006-1138. PMID 17272616
- [Background] Paradisis M, Evans N, Kluckow M, Osborn D. Randomized trial of milrinone versus placebo for prevention of low systemic blood flow in very preterm infants. J Pediatr. 2009 Feb;154(2):189-95. doi: 10.1016/j.jpeds.2008.07.059. Epub 2008 Sep 25. PMID 18822428
- [Background] Bravo MC, Lopez-Ortego P, Sanchez L, Riera J, Madero R, Cabanas F, Pellicer A. Randomized, Placebo-Controlled Trial of Dobutamine for Low Superior Vena Cava Flow in Infants. J Pediatr. 2015 Sep;167(3):572-8.e1-2. doi: 10.1016/j.jpeds.2015.05.037. Epub 2015 Jun 24. PMID 26116470
- [Background] Osborn D, Evans N, Kluckow M. Randomized trial of dobutamine versus dopamine in preterm infants with low systemic blood flow. J Pediatr. 2002 Feb;140(2):183-91. doi: 10.1067/mpd.2002.120834. PMID 11865269
- [Background] Finer NN, Rich W, Wang C, Leone T. Airway obstruction during mask ventilation of very low birth weight infants during neonatal resuscitation. Pediatrics. 2009 Mar;123(3):865-9. doi: 10.1542/peds.2008-0560. PMID 19255015
- [Background] Rich WD, Leone T, Finer NN. Delivery room intervention: improving the outcome. Clin Perinatol. 2010 Mar;37(1):189-202. doi: 10.1016/j.clp.2010.01.011. PMID 20363455
- [Background] Vento M, Aguar M, Leone TA, Finer NN, Gimeno A, Rich W, Saenz P, Escrig R, Brugada M. Using intensive care technology in the delivery room: a new concept for the resuscitation of extremely preterm neonates. Pediatrics. 2008 Nov;122(5):1113-6. doi: 10.1542/peds.2008-1422. No abstract available. PMID 18977992
- [Background] Garey DM, Ward R, Rich W, Heldt G, Leone T, Finer NN. Tidal volume threshold for colorimetric carbon dioxide detectors available for use in neonates. Pediatrics. 2008 Jun;121(6):e1524-7. doi: 10.1542/peds.2007-2708. Epub 2008 May 5. PMID 18458036
- [Background] Leone TA, Lange A, Rich W, Finer NN. Disposable colorimetric carbon dioxide detector use as an indicator of a patent airway during noninvasive mask ventilation. Pediatrics. 2006 Jul;118(1):e202-4. doi: 10.1542/peds.2005-2493. Epub 2006 Jun 26. PMID 16801392
- [Background] Wang CL, Anderson C, Leone TA, Rich W, Govindaswami B, Finer NN. Resuscitation of preterm neonates by using room air or 100% oxygen. Pediatrics. 2008 Jun;121(6):1083-9. doi: 10.1542/peds.2007-1460. PMID 18519476
- [Background] Katheria AC, Harbert MJ, Nagaraj SB, Arnell K, Poeltler DM, Brown MK, Rich W, Hassen KO, Finer N. The Neu-Prem Trial: Neuromonitoring of Brains of Infants Born Preterm During Resuscitation-A Prospective Observational Cohort Study. J Pediatr. 2018 Jul;198:209-213.e3. doi: 10.1016/j.jpeds.2018.02.065. Epub 2018 Apr 18. PMID 29680471
- [Background] Katheria AC, Leone TA, Woelkers D, Garey DM, Rich W, Finer NN. The effects of umbilical cord milking on hemodynamics and neonatal outcomes in premature neonates. J Pediatr. 2014 May;164(5):1045-1050.e1. doi: 10.1016/j.jpeds.2014.01.024. Epub 2014 Feb 20. PMID 24560179
- [Background] Katheria AC, Truong G, Cousins L, Oshiro B, Finer NN. Umbilical Cord Milking Versus Delayed Cord Clamping in Preterm Infants. Pediatrics. 2015 Jul;136(1):61-9. doi: 10.1542/peds.2015-0368. PMID 26122803
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Tataranno ML, Oei JL, Perrone S, Wright IM, Smyth JP, Lui K, Tarnow-Mordi WO, Longini M, Proietti F, Negro S, Saugstad OD, Buonocore G. Resuscitating preterm infants with 100% oxygen is associated with higher oxidative stress than room air. Acta Paediatr. 2015 Aug;104(8):759-65. doi: 10.1111/apa.13039. Epub 2015 Jun 19. PMID 25966608
- [Background] Greisen G. Is near-infrared spectroscopy living up to its promises? Semin Fetal Neonatal Med. 2006 Dec;11(6):498-502. doi: 10.1016/j.siny.2006.07.010. Epub 2006 Sep 7. PMID 16959556
- [Background] Winter J, Kattwinkel J, Chisholm C, Blackman A, Wilson S, Fairchild K. Ventilation of Preterm Infants during Delayed Cord Clamping (VentFirst): A Pilot Study of Feasibility and Safety. Am J Perinatol. 2017 Jan;34(2):111-116. doi: 10.1055/s-0036-1584521. Epub 2016 Jun 15. PMID 27305177
- [Background] Pratesi S, Montano S, Ghirardello S, Mosca F, Boni L, Tofani L, Dani C. Placental Circulation Intact Trial (PCI-T)-Resuscitation With the Placental Circulation Intact vs. Cord Milking for Very Preterm Infants: A Feasibility Study. Front Pediatr. 2018 Nov 27;6:364. doi: 10.3389/fped.2018.00364. eCollection 2018. PMID 30538975
- [Background] Katheria AC, Sorkhi SR, Hassen K, Faksh A, Ghorishi Z, Poeltler D. Acceptability of Bedside Resuscitation With Intact Umbilical Cord to Clinicians and Patients' Families in the United States. Front Pediatr. 2018 Apr 26;6:100. doi: 10.3389/fped.2018.00100. eCollection 2018. PMID 29755962
- [Background] Rabe H, Wacker A, Hulskamp G, Homig-Franz I, Jorch G. Late cord clamping benefits extrauterine adaptation. Pediatric research. 1998;44:454.
- [Background] Nelle, M., Fisher, S., Conze, S. et al. EFFECTS OF LATE CORD CLAMPING ON CIRCULATION IN PREMATURES (VLBWI). Pediatric Research. 1998;44;454
- [Background] Narendra, A., Beckett, C., Aitchison, T. et al. Is it Possible to Promote Placental Transfusion (PTFx) at Preterm Delivery?. Pediatric Research. 1998;44;454
- [Background] Kinmond S, Aitchison TC, Holland BM, Jones JG, Turner TL, Wardrop CA. Umbilical cord clamping and preterm infants: a randomised trial. BMJ. 1993 Jan 16;306(6871):172-5. doi: 10.1136/bmj.306.6871.172. PMID 8443480
- [Background] Ibrahim HM, Krouskop RW, Lewis DF, Dhanireddy R. Placental transfusion: umbilical cord clamping and preterm infants. J Perinatol. 2000 Sep;20(6):351-4. doi: 10.1038/sj.jp.7200408. PMID 11002872
- [Derived] Katheria AC, Ines F, Lee HC, Sollinger C, Vali P, Morales A, Sanjay S, Dorner R, Koo J, Gollin Y, Das A, Poeltler D, Steinhorn R, Finer N, Lakshminrusimha S. Deferred Cord Clamping With High Oxygen in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2025 Sep 1;179(9):971-978. doi: 10.1001/jamapediatrics.2025.2128. PMID 40690234